CLINICAL TRIAL: NCT00088816
Title: Phase II Clinical Study of Preoperative S-1/CDDP Combination Chemotherapy in Patients With Advanced Gastric Cancer
Brief Title: S-1 and Cisplatin Before Surgery in Treating Patients With Stage IV Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyoto University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000368443; KYUH-UHA-GC03-01
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2008-03

CONDITIONS: Gastric Cancer
Keywords: stage IV gastric cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cisplatin; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: tegafur-gimeracil-oteracil potassium
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as S-1 and cisplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Giving combination chemotherapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well giving S-1 together with cisplatin works in treating patients who are undergoing surgery for stage IV gastric cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and feasibility of neoadjuvant chemotherapy comprising S-1 and cisplatin in patients with stage IV gastric adenocarcinoma.
* Determine the overall survival of patients treated with this regimen.

Secondary

* Determine the time to progression and types of initial recurrence in patients treated with this regimen.
* Determine tumor response in patients treated with this regimen.
* Determine mortality and morbidity related to treatment in these patients.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral S-1 on days 1-21 and cisplatin IV over 2 hours on day 8. Treatment repeats every 35 days for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo gastrectomy with lymphadenectomy. Patients resume oral S-1 after surgery.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed gastric adenocarcinoma

  * Stage IV disease meeting 1 of the following staging criteria according to Japanese gastric cancer classification:

    * T4, N2
    * T4, N3
    * P1, CY1
  * CT scan and laparoscopic staging required

PATIENT CHARACTERISTICS:

Age

* 20 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 4,000/mm^3 AND < 12,000/mm^3
* Granulocyte count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin ≤ 1.5 mg/dL

Renal

* Creatinine clearance ≥ 50 mL/min

Pulmonary

* PaO_2 ≥ 70 mm Hg on room air

Other

* Able to swallow oral medication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for gastric cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for gastric cancer

Surgery

* No prior surgery for gastric cancer

Other

* No other prior therapy for gastric cancer

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-04; Primary Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to progression
Tumor response
Death related to treatment
Histological response
Postoperative complications
Surgical/pathological curative resection
Types of initial recurrence
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Seiji Satoh, Study Chair — Kyoto University Hospital
Locations (7):
- Japan (7):
  - Kyoto University Hospital, Kyoto, Kyoto
  - National Hospital Organization - Kyoto Medical Center, Kyoto, Kyoto
  - Kyoto-Katsura Hospital, Kyoto, Kyoto
  - Kitano Hospital, Osaka, Osaka
  - Kansai Denryoku Hospital, Osaka, Osaka
  - Shimane Prefectural Central Hospital, Izumo-shi, Shimane
  - Yamato Municipal Hospital, Yamato City Kanagawa

REFERENCES:
- [Result] Satoh S, Okabe H, Teramukai S, Hasegawa S, Ozaki N, Ueda S, Tsuji A, Sakabayashi S, Fukushima M, Sakai Y. Phase II trial of combined treatment consisting of preoperative S-1 plus cisplatin followed by gastrectomy and postoperative S-1 for stage IV gastric cancer. Gastric Cancer. 2012 Jan;15(1):61-9. doi: 10.1007/s10120-011-0066-9. Epub 2011 Jun 11. PMID 21667134